CLINICAL TRIAL: NCT00531427
Title: Randomized, Double-blind, Placebo-controlled With Open-label Run-in Assessing Efficacy, Tolerability,Safety of BTDS 10 or 20 Compared to Placebo in Opioid-naïve Subjects w/Moderate to Severe, Chronic Pain Due to OA of Knee
Brief Title: Buprenorphine Transdermal System (BTDS) in Subjects w/Mod-sev Osteoarthritis (OA) Chronic Pain of Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3025
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Pain; Osteoarthritis of the Knee
Keywords: Chronic pain,; OA of the knee,; opioid,; transdermal
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Buprenorphine transdermal system 10 and 20 applied for 7-day wear
  Interventions: Drug: Buprenorphine
- 2 (Placebo Comparator): Placebo transdermal system to match BTDS patches, applied for 7-day wear
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — transdermal system 10 and 20 applied for 7-day wear
  Arms: 1
Drug: Placebo — transdermal system (placebo) applied for 7-day wear
  Arms: 2

SUMMARY:
The objective of this study is to determine the analgesic efficacy and safety of Buprenorphine Transdermal System (BTDS) 10 and 20 compared to placebo in opioid-naïve subjects with moderate to severe chronic pain due to osteoarthritis (OA) of the knee. The double-blind treatment intervention duration is 12 weeks, during which time supplemental analgesic medication (immediate-release oxycodone for the first 6 days postrandomization and acetaminophen or ibuprofen for the remainder of the double-blind phase) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic settings for the relief of moderate to severe pain. BTDS is a transdermal system formulation that is designed to deliver a consistent and a steady dose of buprenorphine over a 7-day period with limited blood concentration fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* subjects with moderate to severe chronic osteoarthritis (OA) pain of the knee (lasting several hours daily) as their predominant pain condition,
* clinical diagnosis of OA of the knee 1 year or longer,
* subjects treated within the 14 days prior to screening with nonopioid therapy only, or with therapy including opioids at a dose of < 5 mg oxycodone (or equivalent) per day,
* subjects whose OA knee pain is not adequately controlled with nonopioid analgesic medication and who the investigator feels are appropriate candidates for around-the-clock opioid therapy.

Exclusion Criteria:

* subjects who have had arthroscopy on either knee or hip within 6 months of entering the study or open surgery on either knee or hip within 9 months of entering the study,
* subjects who are allergic to buprenorphine or who have a history of allergies to other opioids,
* subjects who have allergies or other contraindications to transdermal delivery systems or patch adhesives.

Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (83):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Radiant Research, Phoenix Southeast, Chandler, Arizona
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Research Facility, Phoenix, Arizona
  - Research Facility, Anaheim, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Catalina Research Institute, Chino, California
  - Research Facility, Downey, California
  - Research Facility, Foothill Ranch, California
  - Research Facility, Laguna Hills, California
  - Research Facility, Sacramento, California
  - Research Facility, Littleton, Colorado
  - Research Facility, Stamford, Connecticut
  - Coastal Pain Management, Bradenton, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Research Facility, Clearwater, Florida
  - Research Facility, Jupiter, Florida
  - Research Facility, Largo, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Plantation, Florida
  - Research Facility, Royal Palm Hammock, Florida
  - Clinical Research of West Flor, Tampa, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, Venice, Florida
  - Research Facility, West Palm Beach, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Augusta, Georgia
  - AMR Research Associates, Bogart, Georgia
  - Research Facility, Dawsonville, Georgia
  - Research Facility, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Honolulu, Hawaii
  - Rehabilitation Association of IN, Indianapolis, Indiana
  - Research Facility, Overland Park, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Stat-Lab I, Inc., Baton Rouge, Louisiana
  - Research Facility, New Iberia, Louisiana
  - Research Facility, New Orleans, Louisiana
  - Research Facility, Frederick, Maryland
  - Research Facility, Brockton, Massachusetts
  - East Coast Clinical Research, Haverhill, Massachusetts
  - Research Facility, Springfield, Massachusetts
  - Research Facility, Bay City, Michigan
  - Premier Internal Medicine, Biloxi, Mississippi
  - Research Facility, Florissant, Missouri
  - Research Facility, St Louis, Missouri
  - Sports Med Consultants PC, St Louis, Missouri
  - Research Facility, Henderson, Nevada
  - Research Facility, New York, New York
  - Research Facility, Morgantown, North Carolina
  - Research Facility, Winston-Salem, North Carolina
  - Research Facility, Canton, Ohio
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Columbus, Ohio
  - Digestive Endoscopy Center, Dayton, Ohio
  - Research Facility, Dayton, Ohio
  - Research Facility, Middleburg Heights, Ohio
  - Research Facility, Mount Gilead, Ohio
  - Research Facility, Toledo, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Eugene, Oregon
  - Research Facility, Medford, Oregon
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Research Facility, Duncansville, Pennsylvania
  - Oyster Point Family Health Ctr, Lancaster, Pennsylvania
  - Research Facility, Mechanicsburg, Pennsylvania
  - Research Facility, West Reading, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Research Facility, Cranston, Rhode Island
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Arthritis Clinic, PLLC, Jackson, Tennessee
  - Research Facility, Austin, Texas
  - Research Facility, Colleyville, Texas
  - Research Facility, Dallas, Texas
  - Research Facility, Nederland, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Sugarland, Texas
  - Research Facility, Salt Lake City, Utah
  - NDC Medical Center, Norfolk, Virginia
  - Independence Family Medicine, Virginia Beach, Virginia
  - Pacific Northwest Primary Care, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27-Sep-2007 (first patient first visit) to 28-Apr-2009 (last patient last visit) at 83 medical/research sites in US
Pre-assignment Details: Open-label run-in period designed to select those subjects who both tolerated and responded to treatment with BTDS 10 or BTDS 20 (an enriched design). N = 1151 entered the run-in period, and N = 571 completed. One subject was not dosed, therefore N = 570 randomized. N = 3 subjects did not have safety data, therefore N = 567 had double-blind data.
Groups:
- Double-blind BTDS 10 or 20: Buprenorphine transdermal patches (BTDS) 10 or 20 mcg/h applied for 7-day wear
- Double-blind Placebo: Placebo patches to match the BTDS patches applied for 7-day wear
Period: Overall Study
Arm/Group | Double-blind BTDS 10 or 20 | Double-blind Placebo
Started | 282 | 285
Completed | 209 | 191
Not Completed | 73 | 94
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Adverse Event | 44 | 30
Not completed — Lost to Follow-up | 4 | 3
Not completed — Lack of Efficacy | 14 | 39
Not completed — Administrative | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS 10 or 20 | Double-blind Placebo | Total
Number analyzed (Participants) | 282 | 285 | 567
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.75) | 59.1 (9.77) | 59.1 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 181 | 356
  Male | 107 | 104 | 211

OUTCOME MEASURES:

1. Primary Outcome: "Average Pain Over the Last 24 Hours" Score of the Study Knee at Week 12 of the Double Blind Phase.
Description: "Average pain over the last 24 hours" scores of the study knee at week 12 was evaluated on an 11-point scale: 0 = no pain, 10 = worst pain imaginable, recorded daily.
Time Frame: 24 hours (week 12)
Population: The full analysis population is the group of subjects who were randomized and received at least 1 dose of double-blind study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind BTDS 10 or 20 | Double-blind Placebo
Number analyzed (Participants) | 283 | 287
units on a scale
  Screening (Visit 2) | 7.16 (1.340) | 7.06 (1.300)
  Prerandomization (Visit 3) | 2.63 (1.292) | 2.74 (1.186)
  Double-blind Week 12 (Visit 8) | 3.82 (2.644) | 4.22 (2.644)
Statistical Analysis 1: Comparison: Double-blind BTDS 10 or 20 vs Double-blind Placebo; [Week 12 analysis] The null hypothesis was "no group differences." The alternative hypothesis was that BTDS arm was superior to the placebo arm. Pain scale is 11 points (0 = no pain to 10 = pain as bad as you can imagine); Test type: Superiority or Other; p = 0.0853, Mixed Models Analysis; Statistics are based on a mixed effect general linear model; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.80 to 0.05]

2. Secondary Outcome: Mean Daily Number of Tablets of Nonopioid Supplemental Analgesic Used From Week 2 to 12 of the Double-blind Phase.
Description: Subjects were permitted to take sponsor-provided supplemental analgesic medication after week 1 of the double-blind treatment (acetaminophen or ibuprofen).
Time Frame: 10 weeks
Population: Subjects in the full analysis population who took at least 1 dose of supplemental analgesic medication.
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Double-blind BTDS 10 or 20 | Double-blind Placebo
Number analyzed (Participants) | 136 | 154
tablets | 0.701 (0.8139) | 0.740 (0.8566)
Statistical Analysis 1: Comparison: Double-blind BTDS 10 or 20 vs Double-blind Placebo; Categorical analysis P value is based on a Fisher's exact test. Mean daily number of tablets for subjects who took <=1 dose of supplemental analgesia; Test type: Superiority or Other; p = 0.7098, ANCOVA — To control multiplicity and family-wise error rate, a gate-keeping strategy (stepwise approach) was used to evaluate the statistical significance of the secondary variables. If the primary is negative, the secondary P values are descriptive only; with treatment as a factor and screening and pre-randomization mean pain as covariates; Mean Difference (Final Values) = -0.037, 95% CI 2-sided [-0.233 to 0.159]

3. Secondary Outcome: Sleep Disturbance Subscale of the MOS-Sleep Scale at Weeks 4, 8, and 12 of the Double-blind Phase.
Description: The MOS Sleep Scale consists of 12 individual items (4 sleep disturbance, 2 sleep adequacy, 1 quantity of sleep and optimal sleep, 3 somnolence, 1 snoring, and 1 shortness of breath) and takes 5 to 10 minutes to complete. Question 1 is scored on a scale of 1 to 5 ( 1 = 0-15 min to more than 60 min) and Questions 2 to 12 are scored on a scale of 1 to 6 (1 = all of the time to 6 = none of the time. The Sleep Disturbance Subscale score is derived from the scores to Questions 1, 3, 7, and 8 and ranges from 0 to 100, where higher scores indicate greater sleep disturbance.
Time Frame: Weeks 4, 8, and 12 of the double-bind phase
Population: Full Analysis Population (N = 570) consisted of subjects who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind BTDS 10 or 20 | Double-blind Placebo
Number analyzed (Participants) | 283 | 287
units on a scale
  Screening | 49.51 (24.790) | 51.23 (25.945)
  Prerandomization | 23.23 (19.583) | 26.04 (20.822)
  Week 4 | 27.22 (23.086) | 35.08 (25.565)
  Week 8 | 27.46 (23.795) | 34.78 (24.715)
  Week 12 | 29.60 (25.177) | 33.63 (25.606)
Statistical Analysis 1: Comparison: Double-blind BTDS 10 or 20 vs Double-blind Placebo; Weeks 4, 8, 12 analysis The sleep disturbance subscale was analyzed using the mixed effect linear model with fixed effects for treatment (BTDS or placebo) and time (weeks 1, 2, 4, 8, 12) as categorical, screening mean and prerandomization mean value as covariates, and subject as a random effect; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.46, 95% CI 2-sided [-7.44 to -1.48]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) that occurred after the signing of the informed consent up to end of study and 7 days after discontinuation; or Serious AEs occurring up to 30 days following the last study visit were followed until resolution or for up to 30 days.
Description: AEs were obtained through spontaneous reports and subject interview.
Groups:
- Double-blind BTDS: Buprenorphine transdermal patches (BTDS) 10 or 20 mcg/h applied for 7-day wear
- Open-label Run-in Period: The open-label run-in period was designed with duration of time sufficient to select those subjects who both tolerated and responded to treatment with BTDS 10 or BTDS 20 (an enriched design). During this period, subjects were required to discontinue use of all nonstudy drugs used for the treatment of chronic pain and no supplemental analgesic medications were allowed. Subjects who did not tolerate BTDS 5 were discontinued from the study.
Arm/Group | Double-blind BTDS | Double-blind Placebo | Open-label Run-in Period
Serious Adverse Events (participants affected / at risk) | 13/282 | 3/285 | 5/1151
Other Adverse Events (participants affected / at risk) | 108/282 | 53/285 | 520/1151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS (N=282) | Double-blind Placebo (N=285) | Open-label Run-in Period (N=1151)
Arteriosclerosis coronary artery - DEATH (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — DEATH Systematic and nonsystematic assessment
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment One subject experienced bradycardia poststudy
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Hypertensive heart disease - DEATH (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — DEATH Systematic and nonsystematic assessment
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessment
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Noncardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Cardiac procedure complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments One subject experienced acute myocardial infarction poststudy
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Poststudy SAE
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Poststudy SAE
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Poststudy SAE
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Poststudy SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS (N=282) | Double-blind Placebo (N=285) | Open-label Run-in Period (N=1151)
Nausea (Gastrointestinal disorders) | 34 | 14 | 242 — Systematic and nonsystematic assessment
Vomiting (Gastrointestinal disorders) | 19 | 5 | 90 — Systematic and nonsystematic assessment
Constipation (Gastrointestinal disorders) | 19 | 2 | 90 — Systematic and nonsystematic assessment
Application site pruritus (General disorders) | 31 | 18 | 96 — Systematic and nonsystematic assessment
Application site erythema (General disorders) | 21 | 14 | 37 — Systematic and nonsystematic assessment
Application site rash (General disorders) | 16 | 10 | 37 — Systematic and nonsystematic assessment
Fatigue (General disorders) | 7 | 3 | 62 — Systematic and nonsystematic assessment
Dizziness (Nervous system disorders) | 7 | 6 | 132 — Systematic and nonsystematic assessment
Somnolence (Nervous system disorders) | 10 | 5 | 119 — Systematic and nonsystematic assessment
Headache (Nervous system disorders) | 18 | 20 | 93 — Systematic and nonsystematic assessment
Anxiety (Psychiatric disorders) | 16 | 2 | 12 — Systematic and nonsystematic assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days